CLINICAL TRIAL: NCT06568250
Title: Reaching Rural Veterans: Applying Mind-Body Skills for Pain Using a Whole Health Telehealth Intervention
Brief Title: Reaching Rural Veterans: Applying Mind-Body Skills for Pain Using a Whole Health Telehealth Intervention - UG3 Pilot Study
Acronym: RAMP-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Diana J. Burgess, Core Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1UG3NR020929-01 (NIH)
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; mindfulness; complementary therapies; models, biopsychosocial; rural Veterans health
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: RAMP program

INTERVENTIONS:
Behavioral: RAMP program — The RAMP program is a 12-week virtual program consisting of an individual session (50 minutes) with a Whole Health Coach followed by 11 weekly interactive group sessions (90 minutes each) with pre-recorded expert led education videos, mind-body skill training and practice, and facilitated discussions.

SUMMARY:
This project addresses the significant challenge of providing evidence-based non-pharmacologic pain management to rural-dwelling Veterans in the VA healthcare system who have chronic pain. For this preparatory phase (UG3), the investigators will conduct a single-arm pilot study of 40 rural VA patients with chronic pain to assess study feasibility (recruitment and retention), intervention feasibility (fidelity of intervention delivery and participant engagement rates), acceptability, and effectiveness at addressing pre-defined capabilities, opportunities and motivations.

DETAILED DESCRIPTION:
Pain is a complex biophysical, psychological, and social condition and there is a growing evidence base to support several complementary and integrative health (CIH) approaches, which can address pain in a more holistic way. While the VA has become a leader in advancing CIH through its Whole Health Initiative, there remain many barriers, especially for rural patients. This pilot study will assess the feasibility of an innovative telehealth evidence-based intervention for rural VA patients with chronic pain: the Reaching Rural Veterans: Applying Mind-Body Skills for Pain Using a Whole Health Telehealth Intervention (RAMP). RAMP was developed with multiple-levels of VA stakeholders (including rural patients). It was designed to deliver multiple CIH self-management strategies (pain education, mindfulness, pain specific exercises, and cognitive behavioral strategies) in one intervention, to overcome existing barriers to care and improve rural Veterans' pain and important biopsychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veteran participants must be rural dwelling
* Patient's Veterans Affairs (VA) primary care provider is in the Southeast region of the US
* Email address in the VA electronic health record (EHR)
* Report pain at least most days in the past 3 months
* Brief Pain Inventory (BPI) Pain Interference subscale score of 4 or greater
* Willingness and ability to complete study activities including meeting remotely via videoconferencing when program sessions are held

Exclusion Criteria:

* Participation in a prior project conducted by the study team on mindfulness for pain (NCT0456158) or an engagement activities advisor for the current project
* Current enrollment in a research study for pain
* Current enrollment in a similar facilitated, multi-week, multi-modal CIH program
* Severe, poorly controlled psychiatric or substance use disorder (based on chart review using structured checklists, conducted by trained staff who are trained and supervised by a clinical psychologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The RAMP intervention consisted of a 12-week virtual program including an individual session (50 minutes) with a Whole Health Coach followed by 11 weekly interactive group sessions (90 minutes each) with pre-recorded expert led education videos, mind-body skill training and practice, and facilitated discussions.
Period: Overall Study
Arm/Group | Intervention
Started | 40
Completed | 27
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 16
  More than one race | 5
  Unknown or Not Reported | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants Recruited
Description: Number of participants recruited
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 40

2. Primary Outcome: Female Participants Recruited
Description: Percentage of Female Participants Recruited
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 21

3. Primary Outcome: Racial/Ethnic Minoritized Participants Recruited
Description: Percentage of Racial/Ethnic Minoritized Participants Recruited
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 22

4. Primary Outcome: Participant Satisfaction
Description: Percentage of Participants Who Report Being "Somewhat Satisfied" or "Very Satisfied" with the Program on a 7-point Scale
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 29
Participants | 26

5. Primary Outcome: Participant Engagement
Description: Percentage of participants who participated in at least 7 out of 12 sessions either by attending the group session (i.e., synchronous participation) or reporting that they completed any of the session activities on their own (i.e., asynchronous participation)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 27

6. Primary Outcome: Fidelity of Intervention Delivery
Description: Two experts in developing and delivering mind-body interventions for pain independently observed 10% of sessions via videoconference using a structured checklist.
Time Frame: 3 months
Measure: Count of Units; unit: sessions
Units Other Than Participants: sessions
Arm/Group | Intervention
Number analyzed (Participants) | 40
Number analyzed (sessions) | 6
sessions | 6

7. Primary Outcome: Survey Response Rate
Description: Percentage of participants completing post-treatment data collection
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 30

ADVERSE EVENTS:
Time Frame: From consent until 30 days after the last day of study participation (5 months on average).
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT06568250/Prot_SAP_000.pdf